CLINICAL TRIAL: NCT04062357
Title: Effectiveness and Tolerability of Lidocaine 5% Spray in Treatment of Lifelong Premature Ejaculation Patients. A Randomized Single-blind Placebo-controlled Clinical Trial.
Brief Title: Effectiveness and Tolerability of Lidocaine 5% Spray in Treatment of Lifelong Premature Ejaculation Patients.
Acronym: PE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Abu El-Hamd, Assistant Professor of Dermatology, Venereology and Andrology Department, Faculty of Medicine, Sohag University, Egypt., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3/2019
Record Dates: First submitted 2019-08-14; First posted 2019-08-20 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Lidocaine Spray
Keywords: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Group 1 (n₌75); was given on demand lidocaine 5% spray for 8 weeks (One to two applications (1-2 ml) of lidocaine 5% sprays; contain 5 -10 mg of lidocaine, in a metered dose aerosol-delivery system). Group 2 (n₌75); was given placebo in form on demand alcohol spray for 8 weeks (One to two applications (1-2 ml) of alcohol 70% sprays).
Who Masked: Investigator
Masking Description: Patients were randomized evenly categorized into two treatment groups. Patient's distribution in the two groups was according to randomized encoded ballots, and they were unobservant of the type of the topical medications used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine 5% spray (Active Comparator): Group 1 (n₌75); was given on demand lidocaine 5% spray for 8 weeks (One to two applications (1-2 ml) of lidocaine 5% sprays; contain 5 -10 mg of lidocaine, in a metered dose aerosol-delivery system).
  Interventions: Drug: Lidocaine 5% spray
- Placebo (Placebo Comparator): Group 2 (n₌75); was given placebo in form on demand alcohol spray for 8 weeks (One to two applications (1-2 ml) of alcohol 70% sprays).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine 5% spray — Group 1 (n₌75); was given on demand lidocaine 5% spray for 8 weeks (One to two applications (1-2 ml) of lidocaine 5% sprays; contain 5 -10 mg of lidocaine, in a metered dose aerosol-delivery system).
  Arms: lidocaine 5% spray
Other: Placebo — Group 2 (n₌75); was given placebo in form on demand alcohol spray for 8 weeks.
  Arms: Placebo

SUMMARY:
This study aimed to appraise effectiveness and tolerability of lidocaine 5% spray in treatment of patients with premature ejaculation (PE). The current study has been designed as a randomized single-blind placebo-controlled clinical trial. It was done on 150 lifelong PE patients with normal erection. They were randomized evenly categorized into two treatment groups. Group 1 (n₌75); was given on demand lidocaine 5% spray for 8 weeks. Group 2 (n₌75); was given placebo in form on demand alcohol spray for 8 weeks.

DETAILED DESCRIPTION:
This study aimed to appraise effectiveness and tolerability of lidocaine 5% spray in treatment of patients with premature ejaculation (PE). The current study has been designed as a randomized single-blind placebo-controlled clinical trial. It was done on 150 lifelong PE patients with normal erection. They were randomized evenly categorized into two treatment groups. Group 1 (n₌75); was given on demand lidocaine 5% spray for 8 weeks. Group 2 (n₌75); was given placebo in form on demand alcohol spray for 8 weeks. All medications were applied on the glans penis for 10-20 minutes and then cleaned before planed sexual intercourse. Patients were evaluated with Arabic Index of Premature Ejaculation (AIPE) scores, intravaginal ejaculatory latency times (IELTs), and frequency of sexual intercourse before and after treatments.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of lifelong premature ejaculation

Exclusion Criteria:

1. renal or liver diseases,
2. diabetes mellitus,
3. thyroid diseases,
4. chronic prostatitis,
5. neurological diseases
6. allergic reactions to local anesthetics or alcohols.
7. erectil dysfunction

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Arabic Index of Premature Ejaculation Scores | 0-8 weeks after treatment
  Patients were informed to fulfill the questionnaires of Arabic Index of Premature Ejaculation (AIPE).
Intravaginal ejaculatory latency times | 0-8 weeks after treatment
  Patients were informed to sign up intravaginal ejaculatory latency times (IELTs) using stopwatches.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Egypt, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No